CLINICAL TRIAL: NCT00822393
Title: Clinical Phase III Trial to Compare Treosulfan-based Conditioning Therapy With Busulfan-based Reduced-intensity Conditioning (RIC) Prior to Allogeneic Haematopoietic Stem Cell Transplantation in Patients With AML or MDS Considered Ineligible to Standard Conditioning Regimens
Brief Title: Clinical Phase III Trial Treosulfan-based Conditioning Versus Reduced-intensity Conditioning (RIC)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: medac GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MC-FludT.14/L; EudraCT-No.: 2008-002356-18
Record Dates: First submitted 2009-01-13; First posted 2009-01-14 (Estimated); Last update posted 2020-07-30 (Actual); Status verified 2020-07

CONDITIONS: Acute Myeloid Leukemia; Myelodysplastic Syndrome
Keywords: Treosulfan; Busulfan; Conditioning; Allogeneic; Transplantation
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Myelodysplastic Syndromes | interventions — Busulfan; treosulfan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): Busulfan
  Interventions: Drug: Busulfan
- 2 (Experimental): Treosulfan
  Interventions: Drug: Treosulfan

INTERVENTIONS:
Drug: Busulfan — 4 x 0.8 mg/kg/d Intravenous Day -4 and -3
  Arms: 1
Drug: Treosulfan — 10 g/m2/d Intravenous Day -4, -3, -2
  Arms: 2

SUMMARY:
This randomized allogeneic transplantation protocol compares i.v. Treosulfan-based conditioning therapy with reduced intensity i.v. Busulfan-based conditioning in adult AML and MDS patients at increased risk for standard conditioning therapies. The protocol is based on results of previous phase I/II trials evaluating Treosulfan/Fludarabine conditioning prior to allogeneic haematopoietic stem cell transplantation. The reference arm (reduced intensity i.v. Busulfan/Fludarabine) is considered to be accepted medical practice for the study patient population.

DETAILED DESCRIPTION:
To compare efficacy and safety of Treosulfan-based conditioning (test) with i.v. Busulfan-based reduced intensity conditioning (reference).

The statistical aim of the study is to show non-inferiority with respect to:

Event-free survival (EFS) within 2 years after transplantation. Events are defined as relapse of disease, graft failure or death (whatever occurs first).

1. Comparative evaluation of incidence of CTC grade III/IV mucositis/stomatitis between day -6 and day +28
2. Comparative evaluation of overall survival (OS) and cumulative incidence of relapse (RI) as well as non-relapse mortality (NRM) and transplantation-related mortality (TRM)within 2 years after transplantation
3. Comparative evaluation of day +28 conditional cumulative incidence of engraftment
4. Comparative evaluation of day +28 and day +100 incidence of complete donor-type chimerism
5. Comparative evaluation of cumulative incidence of acute and chronic GvHD within 2 years after transplantation
6. Comparative evaluation of incidence of other CTC grade III/IV adverse events between day -6 and day +28

Individual patients will be followed-up for at most 2 years after transplantation. Three confirmatory interim evaluations and one final analysis are planned, which allow to stop the trial as soon as the question of non-inferiority is answered (as outlined below). In addition, post-surveillance with respect to OS and EFS will be conducted one year after transplantation of the last randomised patient.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with acute myeloid leukaemia acc. to WHO, 2008 (AML in complete remission at transplant, i.e. blast counts < 5 % in bone marrow) or myelodysplastic syndrome acc. to WHO, 2008 (MDS with blast counts < 20 % in bone marrow during disease history) indicated for allogeneic haematopoietic progenitor cell transplantation but considered to be at increased risk for standard conditioning therapies according to the following criteria:

   * patients aged ≥ 50 years at transplant and / or
   * patients with a HCT-CI score > 2 [acc. to Sorror et al., 2005]
2. Availability of an HLA-identical sibling donor (MRD) or HLA-identical unrelated donor (MUD). Donor selection is based on molecular high resolution typing (4 digits) of class II alleles of the DRB1 and DQB1 gene loci and molecular (at least) low resolution typing (2 digits) of class I alleles (i.e., antigens) of the HLA- A, B, and C gene loci. In case, no class I and class II completely identical donor (10 out of 10 gene loci) can be identified, one antigen disparity (class I) and/or one allele disparity (class II) between patient and donor are acceptable. Conversely, disparity of two antigens (irrespective of the involved gene loci) cannot be accepted. These definitions for the required degree of histocompatibility apply to the selection of related as well as of unrelated donors.
3. Adult patients of both gender, age 18 - 70 years
4. Karnofsky Index ≥ 60 %
5. Written informed consent
6. Men capable of reproduction and women of childbearing potential must be willing to consent to using a highly effective method of birth control such as condoms, implants, injectables, combined oral contraceptives, IUDs, sexual abstinence or vasectomised partner while on treatment and for at least 6 months thereafter

Exclusion Criteria:

1. Patients with acute promyelocytic leukaemia with t(15;17)(q22;q12) and in CR1
2. Patients considered contra-indicated for allogeneic HSCT due to severe concomitant illness (within three weeks prior to scheduled day -6):

   * patients with severe renal impairment like patients on dialysis or prior renal transplantation or S-creatinine > 3.0 x ULN or calculated creatinine-clearance < 60 ml/min
   * patients with severe pulmonary impairment, DLCOsb (Hb-adjusted)/or FEV1 < 50 % or severe dyspnoea at rest or requiring oxygen supply
   * patients with severe cardiac impairment diagnosed by echocardiography and LVEF < 40 %
   * patients with severe hepatic impairment indicated by hyperbilirubinaemia > 3 x ULN or ALT / AST > 5 x ULN
3. Active malignant involvement of the CNS
4. HIV-positivity, active non-controlled infectious disease under treatment (no decrease of CRP or PCT) including active viral liver infection
5. Previous allogeneic HSCT
6. Pleural effusion or ascites > 1.0 L
7. Pregnancy or lactation
8. Known hypersensitivity to treosulfan, busulfan and/or related ingredients
9. Participation in another experimental drug trial within 4 weeks prior to day -6 of the protocol
10. Non-cooperative behaviour or non-compliance
11. Psychiatric diseases or conditions that might compromise the ability to give informed consent

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 570 (Actual)
Dates: Start 2008-11-24 (Actual); Primary Completion 2018-01-25 (Actual); Study Completion 2018-01-25 (Actual)

PRIMARY OUTCOMES:
Event-free survival (EFS) | within 2 years after transplantation

SECONDARY OUTCOMES:
Comparative evaluation of incidence of CTC grade III/IV mucositis/stomatitis between day -6 and day +28 | between day -6 and day +28

CONTACTS AND LOCATIONS:
Overall Officials: Dietrich W. Beelen, MD, Principal Investigator — University Hospital, Essen
Locations (33):
- Helsinki University Central Hospital, Dept. of Medicine, Helsinki, Finland
- France (2):
  - Centre Hospitalier Lyon Sud, Lyon
  - Hopital Saint-Louis, Paris
- Germany (20):
  - Universitätsklinikum Koeln, Stammzelltransplantation, Cologne
  - Universitätsklinikum Carl Gustav Carus Dresden, Med. Klinik I, Dresden
  - Klinik für Knochenmarktransplantation, Essen
  - Malteser Krankenhaus St. Franziskus-Hospital, Flensburg
  - Universitätsklinikum Freiburg, Freiburg im Breisgau
  - Universitätsmedizin Goettingen, Haematolgie und Onkologie, Göttingen
  - Asklepios Kliniken Hamburg GmbH, Hamburg
  - Universitätsklinikum Heidelberg, Heidelberg
  - Friedrich-Schiller-Universität Jena, Jena
  - Universitätsklinikum Leipzig, Haematologie, internistische Onkologie, Leipzig
  - Johannes-Gutenberg-Universität Mainz, III. Medizinische Klinik, Mainz
  - Klinikum Rechts der Isar der TU München, III. Med. Klinik, München
  - Universitätsklinikum Münster, Münster
  - Klinikum Nürnberg, 5. Medizinische Klinik, Nuremberg
  - Klinikum Oldenburg gGmbH, Oldenburg
  - Klinikum der Universität Regensburg, Regensburg
  - Universität Rostock, Rostock
  - Universität Tübingen, Tübingen
  - Stiftung Deutsche Klinik für Diagnostik, Wiesbaden
  - Klinikum der Universität Würzburg, Würzburg
- St. Istvan and St. Laszlo Hospital of Budapest, Budapest, Hungary
- Italy (7):
  - Azienda Ospedaliera Papa Giovanni XXIII, Bergamo
  - Hematology University of Brescia, Brescia
  - Scientific Institute H. San Raffaele, Milan
  - Ospedale Civile Pescara, Pescara
  - Policlinico Umberto I Univ. La Sapienza, Rome
  - Clinica Ematologica ed Unita di Terapie Cellulari 'Carlo Melzi', Udine
  - Policlinico GB Rossi (Borgo Roma), Div. di Ematologia, Verona
- Poland (2):
  - Medical University of Gdansk, Gdansk
  - Silesian Medical University, Katowice

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Beelen DW, Trenschel R, Stelljes M, Groth C, Masszi T, Remenyi P, Wagner-Drouet EM, Hauptrock B, Dreger P, Luft T, Bethge W, Vogel W, Ciceri F, Peccatori J, Stolzel F, Schetelig J, Junghanss C, Grosse-Thie C, Michallet M, Labussiere-Wallet H, Schaefer-Eckart K, Dressler S, Grigoleit GU, Mielke S, Scheid C, Holtick U, Patriarca F, Medeot M, Rambaldi A, Mico MC, Niederwieser D, Franke GN, Hilgendorf I, Winkelmann NR, Russo D, Socie G, Peffault de Latour R, Holler E, Wolff D, Glass B, Casper J, Wulf G, Menzel H, Basara N, Bieniaszewska M, Stuhler G, Verbeek M, Grass S, Iori AP, Finke J, Benedetti F, Pichlmeier U, Hemmelmann C, Tribanek M, Klein A, Mylius HA, Baumgart J, Dzierzak-Mietla M, Markiewicz M. Treosulfan or busulfan plus fludarabine as conditioning treatment before allogeneic haemopoietic stem cell transplantation for older patients with acute myeloid leukaemia or myelodysplastic syndrome (MC-FludT.14/L): a randomised, non-inferiority, phase 3 trial. Lancet Haematol. 2020 Jan;7(1):e28-e39. doi: 10.1016/S2352-3026(19)30157-7. Epub 2019 Oct 9. PMID 31606445
- See also: Sponsor's homepage — http://www.medac.de